CLINICAL TRIAL: NCT02547740
Title: Structural and Functional Progression of Glaucomatous Damage to the Macula
Brief Title: Macular Damage in Early Glaucoma and Progression
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAAO8502; 1R01EY025253-01 (NIH)
Record Dates: First submitted 2015-09-10; First posted 2015-09-11 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Glaucoma
Keywords: macula; visual fields; optical coherence tomography; glaucoma progression; retinal ganglion cells
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early Glaucomatous Damage: Patients with early functional glaucomatous damage.
- Ophthalmologically Healthy: Healthy subjects that are ophthalmologically normal

SUMMARY:
Glaucoma is the leading cause of irreversible blindness worldwide. This study aims to test a new method that may allow earlier diagnosis of glaucoma and better ways to monitor if it is getting worse. There is scientific evidence that the macula, the central part of the retina, can be involved in very early stages of glaucoma. Glaucomatous damage to the macula is very prevalent and is often missed using conventional clinical tests.

Relatively little is known about progression of early glaucoma damage and its effects on the macula. This project investigates the nature of progressive damage to the macula and proposes new methods to improve accuracy to detect clinically significant progression.The study will evaluate the nature of damage to the macula's structures through OCT imaging and eye function via visual field tests.

DETAILED DESCRIPTION:
There is compelling evidence that glaucomatous damage to the macula occurs even in early stages of the disease. The macula comprises about 30% of all retinal ganglion cells and its information corresponds to over 50% of the visual cortex. However, glaucomatous damage to the macula is often missed in clinical practice. Some of the reasons are:

1. traditional glaucoma knowledge supports that glaucoma is fundamentally a peripheral disease;
2. inherent limitations of conventional clinical tests to detect damage to the macula; and
3. the paucity of large, prospective studies that describe the nature of glaucomatous damage to the macula.

The investigators have published numerous papers in the past two years showing that macular damage is prevalent among patients with early glaucoma if one employs the appropriate tools to assess it, namely 10-2 visual fields and high-resolution optical coherence tomography (OCT). This information comes from a unique prospective cross- sectional database and techniques the investigators developed to produce objective metrics of structure and function.

Now that the investigators understand the cross-sectional nature of macular damage, this proposal aims to:

1. develop a longitudinal database including patients with early glaucoma and healthy controls,
2. to test models that explain progression of macular damage, and
3. to apply new statistical methods combining structural and functional tests which could improve the accuracy to detect progression and shorten the length of clinical trials.

The main hypothesis is that incorporating 10-2 visual field testing and high-resolution OCT scans of the macula to the conventional repertoire of technologies used in clinical practice, in addition to translating recently described statistical methods into softwares that can be used in daily practice, enhances the performance and confidence to detect glaucoma progression.

In Aim 1 the investigators plan to follow healthy subjects and glaucoma patients at regular intervals with 10-2, 24-2 visual fields, and swept source (ss) OCT tests and define metrics of short- and long-term test variability that are needed to differentiate true progression from 'noise'. To date, there is no such database combining these technologies.

In Aim 2 the investigators plan to combine metrics of structure and function from this longitudinal database using two methods: a spatial approach, which will ultimately produce a joint structure-function index using 10-2 and ssOCT data; and a temporal approach, which will employ Bayesian statistics to measure rates of progression using trend analysis. By the end of the study, our contributions to the field should be:

1. to make available a unique and pristine longitudinal database that could be used for other hypotheses testing,
2. to translate techniques recently described in the literature into objective tools to be readily useful in clinical practice, and
3. to mitigate the burdens of progressive loss of central vision in glaucoma.

ELIGIBILITY:
Glaucoma Group:

Inclusion Criteria:

* glaucomatous optic neuropathy (as defined in the American Academy of Ophthalmology Preferred Practice Pattern criteria)

Exclusion Criteria:

* late functional glaucomatous damage
* significant cataract
* previous ocular surgery (aside from uncomplicated cataract extraction with intraocular lens (IOL) implantation and/or trabeculectomy, LASIK or refractive surgeries)
* diabetic retinopathy with macular edema
* vein or artery occlusion
* exudative age-related macular degeneration or geographic atrophy
* macular hole or traction
* amblyopia
* uveitis
* non-open angle glaucoma (e.g. angle closure, traumatic, congenital glaucoma)
* severe myopia or hyperopia (refractive error greater than -6 or +6D, respectively)
* retinal detachment (current or post-surgery)
* retinitis pigmentosa
* significant epiretinal memberane
* significant kerotoconus

Healthy Group:

Inclusion Criteria:

* best corrected visual acuity equal or better than 20/40
* normal biomicroscopy examination
* gonioscopically open angles
* Intraocular Pressure (IOP) lower than 22 mmHg
* normal and reliable 24-2 and 10-2 SAP results

Exclusion Criteria:

* evidence of optic neuropathy
* evidence of clinically significant metabolic diseases (e.g. diabetes and hypotension)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seen in Columbia eye clinics and enrolled in cross-sectional database; Columbia University Medical Center Eye Institute.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Change in 10-2 visual field | Baseline and 3 years
  Evidence of functional glaucomatous damage on the macula as confirmed by visual fields: A slope of 10-2 visual field change faster than -1 dB/year at P<5%
Change in macular ganglion cell thickness | Baseline and 3 years
  Evidence of structural glaucomatous damage on the macula as confirmed by OCT imaging: evidence of macular ganglion cell thickness slope less than -10 microns/year

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Liebmann, MD, Principal Investigator — Columbia University
Locations (1):
- CUIMC Harkness Eye Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hood DC, Tsamis E, Bommakanti NK, Joiner DB, Al-Aswad LA, Blumberg DM, Cioffi GA, Liebmann JM, De Moraes CG. Structure-Function Agreement Is Better Than Commonly Thought in Eyes With Early Glaucoma. Invest Ophthalmol Vis Sci. 2019 Oct 1;60(13):4241-4248. doi: 10.1167/iovs.19-27920. PMID 31618760